CLINICAL TRIAL: NCT04864730
Title: Constitution d'un modèle 3D d'Anatomie Modale de L'Ethmoide Par intégration de Multiples Instances d'Acquisition
Brief Title: Modal Anatomy of the Ethmoid Bone
Acronym: AME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Docteur Patrice GALLET, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI160
Record Dates: First submitted 2020-09-10; First posted 2021-04-29 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2020-09

CONDITIONS: Anatomic Abnormality
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT scans: No intervention Data of voxels will be integrated to the final model
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The creation of a 3D model of modal anatomy of the ethmoid could, like other parts of the body, improve anatomical, radiological and perhaps even surgical learning. Anatomical variations might constitute a "background noise" of the modal anatomy, which can be attenuated by multiplying the instances of acquisitions. The objective of this work is to establish modal anatomy of the ethmoid by the analysis of a large number of CT-scan acquisitions carried out in individuals with no acquired sinus pathology.

DETAILED DESCRIPTION:
Non-interventional descriptive research.

Sinus CTscans (period 2016-2019) will be reviewed from the PACS database of the CHRU of Nancy and selected in individuals without sinus pathology. All CT-scans will be fully anonymized. 26 landmarks will be pointed out to enable :

1. prior images alignment (centering on the median line, realignment rotations then resizing)
2. a mean and median calculation, allowing to establish a mean and median ethmoid model
3. calculation of standard deviations for each voxel The structures obtained in this way (bone, tissue or aerial) will be described anatomically.

ELIGIBILITY:
Retrospective analysis of sinus CT scans images from individuals (period 2016-2019)

Inclusion Criteria:

All individuals (>18 years all) with a sinus CT scan available in the CHRU database

Exclusion Criteria:

inflammatory sinus disease (eg. nasal polyposis, aspergilloma, ...) evolutive sinus tumor anatomical abnormality (e.g. post traumatic, prior sinus surgery, embryologic abnormality...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had a sinus CT-scan during the 2016-2019 period.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Descriptive study of the anatomy of the final 3D model | Through completion of the study: 1 month (The model will be available only at the end of the study, after implementation of all CT-scans)
  Descriptive study
  The study aims to produce the "modal" (generic) model from all the individual sub-models.
  The structures obtained will be described anatomically by ENT experts: the created model will be described in comparison with anatomical data from literature: constant structures (e.g. middle turbinate, inferior turbinate, or orbital wall) will be listed and described (sites of insertion, direction, form), while variations in anatomical structures will be described through the variance (variances of voxels, pooled for each anatomical sub-site) (e.g. anterior ethmoid, sphenoid...). The heat map of voxels' variances will be superposed on the final model.
  No scale/physiological parameter/questionnaire can be used for anatomical description of a single model. Therefore we don't really understand your remark "Please further specify the measurement that will be used (e.g., descriptive name of scale, physiological parameter, questionnaire) to assess this outcome measure."

IPD SHARING:
Plan to Share IPD: No